CLINICAL TRIAL: NCT03324139
Title: Treatment of Intrauterine Growth Restriction With Low Molecular Heparin: Randomized Clinical Trial. Tratamiento Del Crecimiento Intrauterino Restringido Precoz Con Heparina de Bajo Peso Molecular: Ensayo clínico Aleatorizado.
Brief Title: Treatment of Intrauterine Growth Restriction With Low Molecular Heparin.
Acronym: TRACIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Servicio de Asesoría a la Investigación y Logística SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSJD-TRACIP-2017; 2017-001905-33 (EudraCT Number)
Record Dates: First submitted 2017-09-15; First posted 2017-10-27 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Heparin, Low-Molecular-Weight; Heparin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, two-parallel, placebo-controlled, phase III multicenter clinical trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Treatment with low molecular weight Heparin.
  Interventions: Drug: Low molecular weight heparin
- Control Group (Placebo Comparator): Treatment with Placebo.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Low molecular weight heparin — Patients included in this study group will receive 3,500 IU / 0.2 ml / day of Bemiparina sc, from inclusion to delivery (estimated median of 5-6 weeks, with a maximum of 13 weeks).
  Other Names: heparin
  Arms: Study Group
Drug: Placebos — Patients included in this study group will placebo (same presentation as the active drug), from inclusion to delivery (estimated median of 5-6 weeks, with a maximum of 13 weeks).
  Other Names: sodium chloride (0.9%)
  Arms: Control Group

SUMMARY:
TREATMENT OF INTRAUTERINE GROWTH RESTRICTION WITH LOW MOLECULAR WEIGHT HEPARIN.

DETAILED DESCRIPTION:
TREATMENT OF INTRAUTERINE GROWTH RESTRICTION WITH LOW MOLECULAR WEIGHT HEPARIN: RANDOMIZED CLINICAL TRIAL (TRACIP STUDY).

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years.
* Unique gestations
* Diagnosis of early placental intrauterine growth (according to Delphi classification): <32 weeks at diagnosis + Doppler AU with absent / reverse flow or (estimated fetal weight <10 percentile + pulsed Doppler ultrasonography) or (estimated fetal weight <percentile 10 + pulsed uterine artery Doppler).
* Patient giving written informed consent to participate in the study.

Exclusion Criteria:

* Chromosopathies, genetic alterations or fetal malformations.
* Diagnostic treatment with low molecular weight heparins, oral anticoagulants or acetylsalicylic acid prior to inclusion.
* History of heparin-induced thrombocytopenia.
* Active hemorrhage or increased risk of bleeding due to changes in hemostasis.
* Severe hepatic or pancreatic function disorder.
* Organic lesions that may bleed (eg, active peptic ulcer, hemorrhagic stroke, aneurysms, or brain tumors).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 48 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-02-19 (Actual)

PRIMARY OUTCOMES:
Efficacy of low molecular weight heparin in the prolongation of gestation. | 13 weeks maximum
  Measured as gestational age (weeks) at birth (dated by ultrasonography <14 weeks by measurement of caudal skull length).

SECONDARY OUTCOMES:
Efficacy of low molecular weight heparin in reducing neonatal morbidity | 13 weeks maximum
  Measured as the presence of one or more of the following: Perinatal mortality (> 22 weeks of gestation - <28 days postpartum), Significant neonatal morbidity (convulsions, intraventricular haemorrhage> grade III, periventricular leukomalacia, hypoxic-ischemic encephalopathy, abnormal electroencephalogram, necrotizing enterocolitis, acute renal failure (serum creatinine> 1.5 mg / dL) or cardiac failure (requiring inotropic agents), Perinatal mortality (22 weeks to 28 postnatal days), Biomarkers.
Demonstrate that low molecular weight heparin improves the pro-angiogenic and anti-inflammatory profile. | 13 weeks maximum
  Measured as the presence of one or more of the following: mother blood biomarkers (sFlt and PlGF), biomerkers, umbilical cord blood biomarkers (TNF alfa, IL6, IFN gamma, FGF basic, VEGF and PlGF), mRNA in trophoblast.( IL6, INFg, TNF alfa, VEGFA, VEGFB, FGF2 y RQVEGF).
Efficacy of low molecular weight heparin in reducing thrombotic and ischemic placental lesions | 13 weeks maximum
  Measured as the presence of one or more of the following: Intrauterine growth retardation (Neonatal weight below the 10th percentile of our population + umbilical artery pulsatility index during the third trimester (on two separate occasions> 48h) above the 95th percentile), Preeclampsia, Gestational age (weeks) at birth, Premature delivery before 34 weeks of gestation, Urgent cesarean section due to loss of fetal well-being, Neonatal weight, Neonatal acidosis (arterial pH <7.10 + EB> 12mEq / L), Days stay in the Neonatal Intensive Care Unit, mRNA in trophoblast.

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Mazarico, Principal Investigator — Hospital Sant Joan de Deu
Locations (1):
- Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazarico E, Peguero A, Camprubi M, Rovira C, Gomez Roig MD, Oros D, Ibanez-Burillo P, Schoorlemmer J, Masoller N, Tassies MD, Figueras F. Study protocol for a randomised controlled trial: treatment of early intrauterine growth restriction with low molecular weight heparin (TRACIP). BMJ Open. 2018 Oct 23;8(10):e020501. doi: 10.1136/bmjopen-2017-020501. PMID 30355790